CLINICAL TRIAL: NCT02437318
Title: A Phase III Randomized Double-blind, Placebo Controlled Study of Alpelisib in Combination With Fulvestrant for Men and Postmenopausal Women With Hormone Receptor Positive, HER2-negative Advanced Breast Cancer Which Progressed on or After Aromatase Inhibitor Treatment
Brief Title: Study Assessing the Efficacy and Safety of Alpelisib Plus Fulvestrant in Men and Postmenopausal Women With Advanced Breast Cancer Which Progressed on or After Aromatase Inhibitor Treatment.
Acronym: SOLAR-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBYL719C2301; 2015-000340-42 (EudraCT Number)
Record Dates: First submitted 2015-04-22; First posted 2015-05-07 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: BYL719; HR+; HER2-negative; advanced breast cancer; alpelisib; fulvestrant; PI3K; Phase III; ER+; PgR+; men; postmenopausal; aromatase inhibitor; neoplasms
MeSH Terms: conditions — Breast Neoplasms; Multiple Endocrine Neoplasia Type 1; Neoplasms | interventions — Fulvestrant; Alpelisib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fulvestrant + alpelisib (Experimental): Subjects treated with alpelisib (300 mg; oral; once daily) in combination with fulvestrant (500 mg; intramuscular injection on Day 1 and Day 15 of Cycle 1, and then Day 1 of each subsequent 28-day cycle)
  Interventions: Drug: Fulvestrant; Drug: Alpelisib
- Fulvestrant + placebo (Placebo Comparator): Subjects were treated with placebo (300 mg; oral; once daily) in combination with fulvestrant (500 mg; intramuscular injection on Day 1 and Day 15 of Cycle 1, and then Day 1 of each subsequent 28-day cycle)
  Interventions: Drug: Fulvestrant; Drug: Placebo

INTERVENTIONS:
Drug: Fulvestrant — 500 mg of fulvestrant administered via intramuscular injection on Day 1 and Day 15 of Cycle 1, and then Day 1 of each subsequent 28-day cycle
Drug: Alpelisib — 300 mg of alpelisib tablets for oral use administered once daily
  Other Names: BYL719
  Arms: Fulvestrant + alpelisib
Drug: Placebo — 300 mg of placebo tablets for oral use administered once daily
  Arms: Fulvestrant + placebo

SUMMARY:
To determine whether treatment with alpelisib plus fulvestrant prolonged progression-free survival (PFS) compared to fulvestrant and placebo in men and postmenopausal women with hormone receptor positive (HR+), human epidermal growth factor receptor-2 (HER2)-negative advanced breast cancer, who received prior treatment with an aromatase Inhibitor (AI) either as (neo)adjuvant or for advanced disease.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled, international multicenter Phase III study that evaluated the efficacy and safety of treatment with alpelisib plus fulvestrant versus placebo plus fulvestrant in men and postmenopausal women with HR-positive, HER2-negative advanced breast cancer which had progressed on or after AI treatment.

Subjects were allocated to either the PIK3CA mutant or PIK3CA non-mutant cohort, based on central testing of hotspot-mutations in tumor tissue. Subjects with unknown results were not eligible. Within each cohort, subjects were randomized in a 1:1 ratio to receive either alpelisib 300 mg orally once daily (q.d.), in combination with fulvestrant 500 mg intramuscular (i.m.) on Days 1 and 15 of Cycle 1 and Day 1 of a 28-day cycle thereafter, or placebo daily in combination with fulvestrant 500 mg following the same treatment regimen.

Subjects were treated until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason. All subjects who discontinued study treatment were followed for safety, until 30 days after last study treatment administration, except in the case of death, loss to follow-up, or withdrawal of consent.

Subjects who discontinued study treatment for reasons other than disease progression or withdrawal of consent, were followed until disease progression, death, withdrawal of consent, loss to follow-up, or subject/guardian decision (post-treatment efficacy follow-up).

Finally, all subjects were followed for survival after discontinuation of study treatment and tumor evaluations until the subject's death, loss to follow-up, or withdrawal of consent for survival follow-up (post-treatment survival follow-up)

ELIGIBILITY:
Inclusion Criteria:

* If female, the patient was postmenopausal.
* The patient had identified PIK3CA status.
* Patients could be:
* Relapsed with documented evidence of progression while on (neo)adjuvant endocrine therapy or within 12 months from completion of (neo)adjuvant endocrine therapy with no treatment for metastatic disease.
* Relapsed with documented evidence of progression more than 12 months from completion of (neo)adjuvant endocrine therapy and then subsequently progressed with documented evidence of progression while on or after only one line of endocrine therapy for metastatic disease.
* Newly diagnosed with advanced breast cancer, then relapsed with documented evidence of progression while on or after only one line of endocrine therapy.
* The patient had recurrence or progression of the disease during or after AI therapy (i.e., letrozole, anastrozole, exemestane).
* The patient had a histologically and/or cytologically confirmed diagnosis of estrogen-receptor positive breast cancer by a local laboratory and had HER2 negative breast cancer.
* The patient had either measurable disease per RECIST 1.1 criteria or at least one predominantly lytic bone lesion present.
* The patient had adequate bone marrow function.

Exclusion Criteria:

* The patient had symptomatic visceral disease or any disease burden that made the patient ineligible for endocrine therapy per the investigator's best judgment.
* The patient had received prior treatment with chemotherapy (except for neoadjuvant/adjuvant chemotherapy), fulvestrant, any PI3K, mTOR, or AKT inhibitor (pre-treatment with CDK4/6 inhibitors was allowed).
* The patient had inflammatory breast cancer at screening.
* Patients had Child pugh score B or C.
* Patients had an established diagnosis of diabetes mellitus type I or uncontrolled type II.
* The patient had Eastern Cooperative Oncology Group (ECOG) performance status 2 or more.
* The patient had CNS involvement unless he/she was at least 4 weeks from prior therapy completion to starting the study treatment and had a stable CNS tumor at the time of screening and was not receiving steroids and/or enzyme-inducing antiepileptic medications for brain metastases.
* The patient had participated in a prior investigational study within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever was longer.
* The patient had a history of acute pancreatitis within 1 year of screening or a past medical history of chronic pancreatitis.
* The patient relapsed with documented evidence of progression more than 12 months from completion of (neo)adjuvant endocrine therapy with no treatment for metastatic disease.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2015-07-23 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2023-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (184):
- United States (34):
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Beverly Hills Cancer Center, Beverly Hills, California
  - City of Hope National Medical Center, Duarte, California
  - Scripps Green Hospital, La Jolla, California
  - Kaiser Permanent Southern Californi, San Diego, California
  - UCSF, San Francisco, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists-North, St. Petersburg, Florida
  - Rush University Medical Center, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Edward Cancer Center, Naperville, Illinois
  - Fort Wayne Medical Oncology Hematology Inc, Fort Wayne, Indiana
  - St Francis Health Comprehensive Cancer Center, Topeka, Kansas
  - Mercy Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Detroit Clinical Research Center, Owosso, Michigan
  - St Lukes Cancer Institute, Kansas City, Missouri
  - St Vincent Frontier Cancer Center, Billings, Montana
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University Hospitals of Cleveland Seidman Cancer Center, Cleveland, Ohio
  - Good Samaritan Regional Medical Center, Corvallis, Oregon
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Prisma Health Upstate, Greenville, South Carolina
  - Avera Cancer, Sioux Falls, South Dakota
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology PA Dallas Presbyterian Hospital, Dallas, Texas
  - El Paso Texas Oncology, El Paso, Texas
  - Mays Cancer Ctr Uthsa Mdacc, San Antonio, Texas
  - Texas Oncology Northeast Texas, Tyler, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Wenatchee Valley Medical Center, Wenatchee, Washington
- Argentina (4):
  - Novartis Investigative Site, Berazategui, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Rio Negro, Viedma
  - Novartis Investigative Site, La Rioja
- Australia (4):
  - Novartis Investigative Site, Wahroonga, New South Wales
  - Novartis Investigative Site, Wooloongabba, Queensland
  - Novartis Investigative Site, Elizabeth Vale, South Australia
  - Novartis Investigative Site, Melbourne, Victoria
- Austria (2):
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (6):
  - Novartis Investigative Site, Sint-Niklaas, Oost Vlaanderen
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Libramont
  - Novartis Investigative Site, Ottignies
  - Novartis Investigative Site, Verviers
- Brazil (5):
  - Novartis Investigative Site, Natal, Rio Grande do Norte
  - Novartis Investigative Site, Lajeado, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, São José do Rio Preto
  - Novartis Investigative Site, São Paulo
- Bulgaria (3):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (5):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Cambridge, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Québec, Quebec
- Chile (3):
  - Novartis Investigative Site, Temuco, Región de la Araucanía
  - Novartis Investigative Site, Santiago
  - Novartis Investigative Site, Viña del Mar
- Czechia (4):
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Zlín, Czech Republic
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Prague
- France (16):
  - Novartis Investigative Site, Marseille, Bouches Du Rhone
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, La Roche-sur-Yon
  - Novartis Investigative Site, Le Chesnay
  - Novartis Investigative Site, Levallois-Perret
  - Novartis Investigative Site, Lyon 08
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (14):
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Friedrichshafen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Recklinghausen
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Velbert
- Greece (2):
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
- Novartis Investigative Site, Pokfulam, Hong Kong
- Hungary (4):
  - Novartis Investigative Site, Budapest, Pest County
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Szekszárd
- India (3):
  - Novartis Investigative Site, Vijayawada, Andhra Pradesh
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Mumbai
- Israel (5):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (14):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Chieti, CH
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pontedera, PI
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Rionero in Vulture, PZ
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Savona, SV
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Negrar, VR
  - Novartis Investigative Site, Sassari
- Japan (13):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Akashi, Hyōgo
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Kitaadachi-gun, Saitama
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Minato Ku, Tokyo
  - Novartis Investigative Site, Kagoshima
  - Novartis Investigative Site, Kumamoto
- Lebanon (3):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
  - Novartis Investigative Site, Saida
- Mexico (2):
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, San Luis Potosí City
- Netherlands (2):
  - Novartis Investigative Site, Venray, CE
  - Novartis Investigative Site, Terneuzen
- Peru (3):
  - Novartis Investigative Site, San Borja, Lima region
  - Novartis Investigative Site, Surquillo, Lima region
  - Novartis Investigative Site, Lima
- Romania (3):
  - Novartis Investigative Site, Floreşti, Cluj
  - Novartis Investigative Site, Craiova, Dolj
  - Novartis Investigative Site, Iași
- Russia (3):
  - Novartis Investigative Site, Arkhangelsk
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
- South Korea (3):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Seoul
- Spain (15):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Jerez de la Frontera, Cadiz
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Badajoz, Extremadura
  - Novartis Investigative Site, Cáceres, Extremadura
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Castellon, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Sweden (3):
  - Novartis Investigative Site, Gävle
  - Novartis Investigative Site, Örebro
  - Novartis Investigative Site, Västerås
- Novartis Investigative Site, Taipei, Taiwan
- Novartis Investigative Site, Bangkok, Thailand
- United Kingdom (3):
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Borrego MR, Lu YS, Reyes-Cosmelli F, Park YH, Yamashita T, Chiu J, Airoldi M, Turner N, Fein L, Ghaznawi F, Singh J, Pantoja K, Schnell C, Akdere M, Chia S. SGLT2 inhibition improves PI3Kalpha inhibitor-induced hyperglycemia: findings from preclinical animal models and from patients in the BYLieve and SOLAR-1 trials. Breast Cancer Res Treat. 2024 Nov;208(1):111-121. doi: 10.1007/s10549-024-07405-8. Epub 2024 Aug 23. PMID 39177931
- [Derived] Rodon J, Demanse D, Rugo HS, Burris HA, Simo R, Farooki A, Wellons MF, Andre F, Hu H, Vuina D, Quadt C, Juric D. A risk analysis of alpelisib-induced hyperglycemia in patients with advanced solid tumors and breast cancer. Breast Cancer Res. 2024 Mar 4;26(1):36. doi: 10.1186/s13058-024-01773-1. PMID 38439079
- [Derived] Ciruelos EM, Rugo HS, Mayer IA, Levy C, Forget F, Delgado Mingorance JI, Safra T, Masuda N, Park YH, Juric D, Conte P, Campone M, Loibl S, Iwata H, Zhou X, Park J, Ridolfi A, Lorenzo I, Andre F. Patient-Reported Outcomes in Patients With PIK3CA-Mutated Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer From SOLAR-1. J Clin Oncol. 2021 Jun 20;39(18):2005-2015. doi: 10.1200/JCO.20.01139. Epub 2021 Mar 29. PMID 33780274
- [Derived] Andre F, Ciruelos EM, Juric D, Loibl S, Campone M, Mayer IA, Rubovszky G, Yamashita T, Kaufman B, Lu YS, Inoue K, Papai Z, Takahashi M, Ghaznawi F, Mills D, Kaper M, Miller M, Conte PF, Iwata H, Rugo HS. Alpelisib plus fulvestrant for PIK3CA-mutated, hormone receptor-positive, human epidermal growth factor receptor-2-negative advanced breast cancer: final overall survival results from SOLAR-1. Ann Oncol. 2021 Feb;32(2):208-217. doi: 10.1016/j.annonc.2020.11.011. Epub 2020 Nov 25. PMID 33246021
- [Derived] Rugo HS, Andre F, Yamashita T, Cerda H, Toledano I, Stemmer SM, Jurado JC, Juric D, Mayer I, Ciruelos EM, Iwata H, Conte P, Campone M, Wilke C, Mills D, Lteif A, Miller M, Gaudenzi F, Loibl S. Time course and management of key adverse events during the randomized phase III SOLAR-1 study of PI3K inhibitor alpelisib plus fulvestrant in patients with HR-positive advanced breast cancer. Ann Oncol. 2020 Aug;31(8):1001-1010. doi: 10.1016/j.annonc.2020.05.001. Epub 2020 May 13. PMID 32416251
- [Derived] Andre F, Ciruelos E, Rubovszky G, Campone M, Loibl S, Rugo HS, Iwata H, Conte P, Mayer IA, Kaufman B, Yamashita T, Lu YS, Inoue K, Takahashi M, Papai Z, Longin AS, Mills D, Wilke C, Hirawat S, Juric D; SOLAR-1 Study Group. Alpelisib for PIK3CA-Mutated, Hormone Receptor-Positive Advanced Breast Cancer. N Engl J Med. 2019 May 16;380(20):1929-1940. doi: 10.1056/NEJMoa1813904. PMID 31091374

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in 198 centers across 31 countries
Pre-assignment Details: One subject in the PIK3CA mutant cohort, who was randomized to the placebo + fulvestrant arm, did not receive study treatment due to a protocol deviation.
Groups:
- Alpelisib + Fulvestrant: Subjects treated with alpelisib (300 mg; oral; once daily) in combination with fulvestrant (500 mg; intramuscular injection on Day 1 and Day 15 of Cycle 1, and then Day 1 of each subsequent 28-day cycle)
- Placebo + Fulvestrant: Subjects treated with placebo (300 mg; oral; once daily) in combination with fulvestrant (500 mg; intramuscular injection on Day 1 and Day 15 of Cycle 1, and then Day 1 of each subsequent 28-day cycle)
Period: Overall Study
Arm/Group | Alpelisib + Fulvestrant | Placebo + Fulvestrant
Started | 284 | 288
Treated | 284 | 287
PIK3CA Mutant Cohort by Tumor Tissue (Subjects with advanced breast cancer with a PIK3CA mutation based on central testing of hotspot-mutations in tumor tissue) | 169 | 172
PIK3CA Non-mutant Cohort by Tumor Tissue (Subjects with advanced breast cancer without a PIK3CA mutation based on central testing of hotspot-mutations in tumor tissue) | 115 | 116
PIK3CA Mutant Cohort by ctDNA (Subjects with advanced breast cancer with a PIK3CA mutation measured in ctDNA) | 92 | 94
PIK3CA Non-mutant Cohort by ctDNA (Subjects with advanced breast cancer without a PIK3CA mutation measured in ctDNA) | 181 | 182
Completed | 0 | 0
Not Completed | 284 | 288
Not completed — Progressive disease | 207 | 240
Not completed — Subject/guardian decision | 24 | 11
Not completed — Physician Decision | 29 | 22
Not completed — Adverse Event | 14 | 4
Not completed — Death | 4 | 4
Not completed — Protocol deviation | 5 | 7
Not completed — Sponsor decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alpelisib + Fulvestrant | Placebo + Fulvestrant | Total
Number analyzed (Participants) | 284 | 288 | 572
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.6 (9.74) | 63.3 (10.26) | 63.0 (10.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 283 | 288 | 571
  Male | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 199 | 178 | 377
  Asian | 59 | 66 | 125
  Black or African American | 2 | 6 | 8
  American Indian or Alaska | 1 | 4 | 5
  Other | 9 | 17 | 26
  Unknown | 14 | 17 | 31

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Per Investigator Assessment in the PIK3CA Mutant Cohort
Description: PFS was defined as the time from the date of randomization to the date of the first documented progression or death due to any cause. PFS was assessed via a local radiology assessment according to RECIST 1.1. If a patient did not have an event, PFS was censored at the date of last adequate tumor assessment.
  The PFS distribution was estimated using Kaplan-Meier methodology. Progression was defined as at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Once approximately 243 PFS events in the PIK3CA mutant cohort had been observed, up to 33.3 months
Population: All subjects with a PIK3CA mutation (based on central testing of hotspot-mutations in tumor tissue) who were randomized to study treatment
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- PIK3CA Mutant Cohort by Tumor Tissue: Alpelisib + Fulvestrant: Subjects with advanced breast cancer with a PIK3CA mutation (based on central testing of hotspot-mutations in tumor tissue) treated with alpelisib (300 mg; oral; once daily) in combination with fulvestrant (500 mg; intramuscular injection on Day 1 and Day 15 of Cycle 1, and then Day 1 of each subsequent 28-day cycle)
- PIK3CA Mutant Cohort by Tumor Tissue: Placebo + Fulvestrant: Subjects with advanced breast cancer with a PIK3CA mutation (based on central testing of hotspot-mutations in tumor tissue) treated with placebo (300 mg; oral; once daily) in combination with fulvestrant (500 mg; intramuscular injection on Day 1 and Day 15 of Cycle 1, and then Day 1 of each subsequent 28-day cycle)
Arm/Group | PIK3CA Mutant Cohort by Tumor Tissue: Alpelisib + Fulvestrant | PIK3CA Mutant Cohort by Tumor Tissue: Placebo + Fulvestrant
Number analyzed (Participants) | 169 | 172
Months | 11.0 [7.49 to 14.52] | 5.7 [3.65 to 7.36]
Statistical Analysis 1: Comparison: PIK3CA Mutant Cohort by Tumor Tissue: Alpelisib + Fulvestrant vs PIK3CA Mutant Cohort by Tumor Tissue: Placebo + Fulvestrant; Test type: Superiority; p = 0.00065, Log Rank — (one-sided); Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.50 to 0.85]

2. Secondary Outcome: Overall Survival (OS) in the PIK3CA Mutant Cohort
Description: OS was defined as the time from date of randomization to date of death due to any cause. If a patient was not known to have died, survival was censored at the date of last known date patient alive.
  The OS distribution was estimated using Kaplan-Meier methodology.
Time Frame: Once approximately 178 deaths in the PIK3CA mutant cohort had been observed, up to 55.7 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PIK3CA Mutant Cohort by Tumor Tissue: Alpelisib + Fulvestrant | PIK3CA Mutant Cohort by Tumor Tissue: Placebo + Fulvestrant
Number analyzed (Participants) | 169 | 172
Months | 39.3 [34.10 to 44.85] | 31.4 [26.78 to 41.30]

3. Secondary Outcome: PFS Per Investigator Assessment in the PIK3CA Non-mutant Cohort
Description: as for outcome 1
Time Frame: Up to 56.4 months
Population: All subjects without a PIK3CA mutation (based on central testing of hotspot-mutations in tumor tissue) who were randomized to study treatment
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- PIK3CA Non-mutant Cohort by Tumor Tissue: Alpelisib + Fulvestrant: Subjects with advanced breast cancer without a PIK3CA mutation (based on central testing of hotspot-mutations in tumor tissue) treated with alpelisib (300 mg; oral; once daily) in combination with fulvestrant (500 mg; intramuscular injection on Day 1 and Day 15 of Cycle 1, and then Day 1 of each subsequent 28-day cycle)
- PIK3CA Non-mutant Cohort by Tumor Tissue: Placebo + Fulvestrant: Subjects with advanced breast cancer without a PIK3CA mutation (based on central testing of hotspot-mutations in tumor tissue) treated with placebo (300 mg; oral; once daily) in combination with fulvestrant (500 mg; intramuscular injection on Day 1 and Day 15 of Cycle 1, and then Day 1 of each subsequent 28-day cycle)
Arm/Group | PIK3CA Non-mutant Cohort by Tumor Tissue: Alpelisib + Fulvestrant | PIK3CA Non-mutant Cohort by Tumor Tissue: Placebo + Fulvestrant
Number analyzed (Participants) | 115 | 116
Months | 7.43 [5.55 to 10.84] | 7.23 [5.06 to 9.17]

4. Secondary Outcome: OS in the PIK3CA Non-mutant Cohort
Description: as for outcome 2
Time Frame: Up to 56.4 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PIK3CA Non-mutant Cohort by Tumor Tissue: Alpelisib + Fulvestrant | PIK3CA Non-mutant Cohort by Tumor Tissue: Placebo + Fulvestrant
Number analyzed (Participants) | 115 | 116
Months | 37.29 [27.89 to 45.47] | 34.30 [26.81 to 39.03]

5. Secondary Outcome: Overall Response Rate (ORR) Per Investigator Assessment
Description: ORR was defined as the percentage of patients with best overall response of complete response (CR) or partial response (PR) based on local investigator's assessment according to RECIST 1.1.
  CR: Disappearance of all non-nodal target and non-target lesions. In addition, any pathological lymph nodes assigned as target and non-target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to 56.4 months
Population: All subjects who were randomized to study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PIK3CA Mutant Cohort by Tumor Tissue: Alpelisib + Fulvestrant | PIK3CA Mutant Cohort by Tumor Tissue: Placebo + Fulvestrant | PIK3CA Non-mutant Cohort by Tumor Tissue: Alpelisib + Fulvestrant | PIK3CA Non-mutant Cohort by Tumor Tissue: Placebo + Fulvestrant
Number analyzed (Participants) | 169 | 172 | 115 | 116
Percentage of participants | 26.6 [20.1 to 34.0] | 13.4 [8.7 to 19.4] | 20.9 [13.9 to 29.4] | 12.9 [7.4 to 20.4]

6. Secondary Outcome: Clinical Benefit Rate (CBR) Per Investigator Assessment
Description: Clinical benefit rate was defined as the percentage of patients with a best overall response of CR or PR or stable disease (SD) or Non-CR/Non-PD lasting more than 24 weeks based on local investigator assessment according to RECIST 1.1.
  CR: Disappearance of all non-nodal target and non-target lesions. In addition, any pathological lymph nodes assigned as target and non-target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Up to 56.4 months
Population: All subjects who were randomized to study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PIK3CA Mutant Cohort by Tumor Tissue: Alpelisib + Fulvestrant | PIK3CA Mutant Cohort by Tumor Tissue: Placebo + Fulvestrant | PIK3CA Non-mutant Cohort by Tumor Tissue: Alpelisib + Fulvestrant | PIK3CA Non-mutant Cohort by Tumor Tissue: Placebo + Fulvestrant
Number analyzed (Participants) | 169 | 172 | 115 | 116
Percentage of participants | 61.5 [53.8 to 68.9] | 44.8 [37.2 to 52.5] | 53.9 [44.4 to 63.2] | 49.1 [39.7 to 58.6]

7. Secondary Outcome: Time to Definitive Deterioration of Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) Score From Baseline
Description: ECOG PS categorized patients based on their ability to perform daily activities and self-care, with scores ranging from 0 to 5. A score of 0 indicated no restrictions in activity, while higher scores indicated increasing limitations. Time to definitive deterioration of ECOG PS by one score was defined as the time from the date of randomization to the date of the event, defined as experiencing at least one score lower than the baseline. A deterioration was considered definitive if no improvements in the ECOG PS were observed at a subsequent time. The Kaplan-Meier method was used to estimate the distribution. Patients receiving any further therapy prior to definitive worsening were censored at their date of last assessment prior to start of therapy. Patients that had not worsened at the data cutoff point were censored at the date of last assessment.
Time Frame: From baseline up to 56.4 months
Population: All subjects who were randomized to study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PIK3CA Mutant Cohort by Tumor Tissue: Alpelisib + Fulvestrant | PIK3CA Mutant Cohort by Tumor Tissue: Placebo + Fulvestrant | PIK3CA Non-mutant Cohort by Tumor Tissue: Alpelisib + Fulvestrant | PIK3CA Non-mutant Cohort by Tumor Tissue: Placebo + Fulvestrant
Number analyzed (Participants) | 169 | 172 | 115 | 116
Months | 34.07 [26.32 to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [22.11 to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [13.83 to NA] — NA: Not estimable due to the insufficient number of participants with events | 40.44 [18.46 to 47.21]

8. Secondary Outcome: Time to 10% Deterioration in the Global Health Status (GHS) /Quality of Life (QOL) Scale Score of the European Organization for Research and Treatment of Cancer's Core Quality of Life Questionnaire (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 is a questionnaire that includes 5 functional scales, 3 symptom scales, 1 GHS/QoL scale, and 6 single items. GHS/QoL scale score ranges between 0 and 100. A high score for GHS/QoL represents better functioning or QoL.The time to definitive 10% deterioration was defined as the time from the date of randomization to the date of event, which was defined as at least 10% relative to baseline worsening of the GHS/QoL score (without further improvement above the threshold) or death due to any cause. The Kaplan-Meier method was used to estimate the distribution. If a patient had not had an event, time to deterioration was censored at the date of the last adequate QoL evaluation.
Time Frame: From baseline up to 55.7 months
Population: All subjects who were randomized to study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PIK3CA Mutant Cohort by Tumor Tissue: Alpelisib + Fulvestrant | PIK3CA Mutant Cohort by Tumor Tissue: Placebo + Fulvestrant | PIK3CA Non-mutant Cohort by Tumor Tissue: Alpelisib + Fulvestrant | PIK3CA Non-mutant Cohort by Tumor Tissue: Placebo + Fulvestrant
Number analyzed (Participants) | 169 | 172 | 115 | 116
Months | 18.14 [14.55 to 28.68] | 19.98 [11.50 to 25.59] | 7.39 [5.62 to NA] — NA: not estimable due to the insufficient number of participants with events | 9.23 [3.94 to 13.17]

9. Secondary Outcome: Change From Baseline in the GHS/QOL Scale Score of the EORTC QLQ-C30
Description: The EORTC QLQ-C30 is a questionnaire that includes 5 functional scales, 3 symptom scales, 1 GHS/QoL scale, and 6 single items. GHS/QoL scale score ranges between 0 and 100. A high score for GHS/QoL represents better functioning or QoL.The change from baseline in the GHS/QoL score was assessed. A positive change from baseline indicated improvement.
  For each cohort, this analysis only included assessments up to the time point where there were at least 10 patients on each of the 2 treatment groups.
Time Frame: Baseline, every 8 weeks after randomization during the first 18 months and thereafter every 12 weeks, up to 120 weeks.
Population: Randomized participants with baseline scores and at least one non-missing post-baseline assessment. Number analyzed refers to the number of participants with an evaluable value at the specified time point
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | PIK3CA Mutant Cohort by Tumor Tissue: Alpelisib + Fulvestrant | PIK3CA Mutant Cohort by Tumor Tissue: Placebo + Fulvestrant | PIK3CA Non-mutant Cohort by Tumor Tissue: Alpelisib + Fulvestrant | PIK3CA Non-mutant Cohort by Tumor Tissue: Placebo + Fulvestrant
Number analyzed (Participants) | 142 | 140 | 98 | 92
Score on a Scale
  Week 8 | -2.477 (2.286) | -0.369 (2.324) | 1.524 (2.578) | 2.698 (2.601)
  Week 16: number analyzed (Participants) | 124 | 107 | 66 | 66
  Week 16 | -1.796 (2.349) | -2.685 (2.455) | 2.866 (2.809) | 1.700 (2.835)
  Week 24: number analyzed (Participants) | 105 | 81 | 46 | 34
  Week 24 | -3.010 (2.415) | -0.337 (2.587) | 1.383 (3.087) | 4.909 (3.385)
  Week 32: number analyzed (Participants) | 86 | 73 | 32 | 25
  Week 32 | -2.802 (2.519) | -0.891 (2.646) | 1.063 (3.420) | 4.345 (3.731)
  Week 40: number analyzed (Participants) | 75 | 62 | 12 | 20
  Week 40 | -2.815 (2.581) | -1.854 (2.739) | 13.232 (4.783) | 4.923 (4.003)
  Week 48: number analyzed (Participants) | 69 | 51 | 0 | 0
  Week 48 | -3.635 (2.621) | -1.460 (2.853) |  |
  Week 56: number analyzed (Participants) | 59 | 45 | 0 | 0
  Week 56 | -1.617 (2.701) | 0.248 (2.935) |  |
  Week 64: number analyzed (Participants) | 47 | 42 | 0 | 0
  Week 64 | -1.937 (2.835) | -1.979 (2.984) |  |
  Week 72: number analyzed (Participants) | 48 | 36 | 0 | 0
  Week 72 | -2.525 (2.823) | -1.526 (3.098) |  |
  Week 84: number analyzed (Participants) | 40 | 34 | 0 | 0
  Week 84 | -1.135 (2.958) | -1.495 (3.143) |  |
  Week 96: number analyzed (Participants) | 35 | 25 | 0 | 0
  Week 96 | -3.869 (3.054) | -3.581 (3.423) |  |
  Week 108: number analyzed (Participants) | 26 | 21 | 0 | 0
  Week 108 | -2.158 (3.328) | -2.068 (3.609) |  |
  Week 120: number analyzed (Participants) | 28 | 17 | 0 | 0
  Week 120 | -2.928 (3.251) | -2.593 (3.868) |  |

10. Secondary Outcome: Trough Plasma Concentration of Alpelisib
Description: Pre-dose plasma concentrations of alpelisib were assessed. Only participants randomized to the alpelisib + fulvestrant arm were included in this analysis.
Time Frame: Day 8 and Day 15 of Cycle 1, then Day 1 of Cycles 2, 4, 6 and 8. Cycle = 28 days
Population: Participants who received at least one dose of alpelisib and provided at least one evaluable trough plasma concentration for alpelisib at the specified time points
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)/ milliliter (mL)
Groups:
- Alpelisib + Fulvestrant: Subjects with advanced breast cancer with or without a PIK3CA mutation treated with alpelisib (300 mg; oral; once daily) in combination with fulvestrant (500 mg; intramuscular injection on Day 1 and Day 15 of Cycle 1, and then Day 1 of each subsequent 28-day cycle)
Arm/Group | Alpelisib + Fulvestrant
Number analyzed (Participants) | 96
nanogram (ng)/ milliliter (mL)
  Cycle 1 Day 8 | 424 (41.1)
  Cycle 1 Day 15: number analyzed (Participants) | 64
  Cycle 1 Day 15 | 468 (57.6)
  Cycle 2 Day 1: number analyzed (Participants) | 92
  Cycle 2 Day 1 | 436 (53.4)
  Cycle 4 Day 1: number analyzed (Participants) | 61
  Cycle 4 Day 1 | 458 (69.4)
  Cycle 6 Day 1: number analyzed (Participants) | 44
  Cycle 6 Day 1 | 418 (57.1)
  Cycle 8 Day 1: number analyzed (Participants) | 36
  Cycle 8 Day 1 | 469 (58.3)

11. Secondary Outcome: Trough Plasma Concentration of Fulvestrant
Description: Pre-dose plasma concentrations of fulvestrant were assessed.
Time Frame: Day 15 of Cycle 1, then Day 1 of Cycles 2, 4, 6 and 8. Cycle = 28 days
Population: Participants who received at least one dose of fulvestrant and provided at least one evaluable trough plasma concentration for fulvestrant at the specified time points
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)/ milliliter (mL)
Groups:
- Placebo + Fulvestrant: Subjects with advanced breast cancer with or without a PIK3CA mutation treated with placebo (300 mg; oral; once daily) in combination with fulvestrant (500 mg; intramuscular injection on Day 1 and Day 15 of Cycle 1, and then Day 1 of each subsequent 28-day cycle)
Arm/Group | Alpelisib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 124 | 124
nanogram (ng)/ milliliter (mL)
  Cycle 1 Day 15: number analyzed (Participants) | 106 | 124
  Cycle 1 Day 15 | 10.8 (43.5) | 10.3 (51.0)
  Cycle 2 Day 1: number analyzed (Participants) | 89 | 98
  Cycle 2 Day 1 | 14.0 (39.7) | 14.7 (41.2)
  Cycle 4 Day 1: number analyzed (Participants) | 91 | 74
  Cycle 4 Day 1 | 11.5 (32.2) | 12.2 (29.8)
  Cycle 6 Day 1: number analyzed (Participants) | 124 | 98
  Cycle 6 Day 1 | 12.6 (30.5) | 14.0 (24.2)
  Cycle 8 Day 1: number analyzed (Participants) | 52 | 55
  Cycle 8 Day 1 | 13.5 (35.2) | 14.7 (23.2)

12. Secondary Outcome: PFS Per Investigator Criteria in Subjects With PIK3CA Mutation Status Measured in ctDNA at Baseline
Description: PFS was defined as the time from the date of randomization to the date of the first documented progression or death due to any cause. PFS was assessed via a local radiology assessment according to RECIST 1.1. If a patient did not have an event, PFS was censored at the date of last adequate tumor assessment. The PFS distribution was estimated using Kaplan-Meier methodology.
  Subjects were analyzed according to the PIK3CA mutation status (mutant or non-mutant) as identified using plasma ctDNA.
  Progression was defined as at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From baseline up to 56.4 months
Population: Subjects who were randomized to study treatment with an evaluable mutation status by ctDNA at baseline
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- PIK3CA Mutant Determined by ctDNA: Alpelisib + Fulvestrant: Subjects with advanced breast cancer with a PIK3CA mutation (measured in ctDNA) treated with alpelisib (300 mg; oral; once daily) in combination with fulvestrant (500 mg; intramuscular injection on Day 1 and Day 15 of Cycle 1, and then Day 1 of each subsequent 28-day cycle)
- PIK3CA Mutant Determined by ctDNA: Placebo + Fulvestrant: Subjects with advanced breast cancer with a PIK3CA mutation (measured in ctDNA) treated with placebo (300 mg; oral; once daily) in combination with fulvestrant (500 mg; intramuscular injection on Day 1 and Day 15 of Cycle 1, and then Day 1 of each subsequent 28-day cycle)
- PIK3CA Non-mutant Determined by ctDNA: Alpelisib + Fulvestrant: Subjects with advanced breast cancer without a PIK3CA mutation (measured in ctDNA) treated with alpelisib (300 mg; oral; once daily) in combination with fulvestrant (500 mg; intramuscular injection on Day 1 and Day 15 of Cycle 1, and then Day 1 of each subsequent 28-day cycle)
- PIK3CA Non-mutant Determined by ctDNA: Placebo + Fulvestrant: Subjects with advanced breast cancer without a PIK3CA mutation (measured in ctDNA) treated with placebo (300 mg; oral; once daily) in combination with fulvestrant (500 mg; intramuscular injection on Day 1 and Day 15 of Cycle 1, and then Day 1 of each subsequent 28-day cycle)
Arm/Group | PIK3CA Mutant Determined by ctDNA: Alpelisib + Fulvestrant | PIK3CA Mutant Determined by ctDNA: Placebo + Fulvestrant | PIK3CA Non-mutant Determined by ctDNA: Alpelisib + Fulvestrant | PIK3CA Non-mutant Determined by ctDNA: Placebo + Fulvestrant
Number analyzed (Participants) | 92 | 94 | 181 | 182
Months | 10.9 [7.03 to 15.28] | 3.7 [2.27 to 6.11] | 9.0 [7.23 to 11.01] | 7.4 [5.55 to 9.20]

13. Post Hoc Outcome: All Collected Deaths
Description: Pre-treatment deaths were collected from randomization to the day before first dose of study medication.
  On-treatment deaths were collected from start of treatment to 30 days after last dose of study medication.
  Post-treatment survival follow-up deaths were collected from day 31 after last dose of study treatment to end of study.
Time Frame: Pre-treatment: Up to 35 days. On-treatment: Up to approx. 6.5 years. Post-treatment survival follow-up: Up to approx. 6.5 years
Population: All subjects who were randomized to study treatment.
Measure: Number; unit: Participants
Arm/Group | Alpelisib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 284 | 288
Participants
  Pre-treatment | 0 | 0
  On-treatment: number analyzed (Participants) | 284 | 287
  On-treatment | 9 | 12
  Post-treatment survival follow-up: number analyzed (Participants) | 275 | 275
  Post-treatment survival follow-up | 151 | 156
  All deaths | 160 | 168

14. Other Pre Specified Outcome: Updated PFS Per Investigator Assessment in the PIK3CA Mutant Cohort (Longer Follow-up)
Description: PFS was defined as the time from the date of randomization to the date of the first documented progression or death due to any cause. PFS was assessed via a local radiology assessment according to RECIST 1.1. If a patient did not have an event, PFS was censored at the date of last adequate tumor assessment.
  The PFS distribution was estimated using Kaplan-Meier methodology. This analysis was conducted at the time of the final OS analysis (when approximately 178 deaths in the PIK3CA mutant cohort had been achieved) and includes a longer follow-up time.
  Progression was defined as at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to 55.7 months
Population: All subjects with a PIK3CA mutation who were randomized to study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PIK3CA Mutant Cohort by Tumor Tissue: Alpelisib + Fulvestrant | PIK3CA Mutant Cohort by Tumor Tissue: Placebo + Fulvestrant
Number analyzed (Participants) | 169 | 172
Months | 10.97 [7.49 to 14.52] | 5.65 [3.65 to 7.36]

ADVERSE EVENTS:
Time Frame: All-cause mortality: from randomization up to approx. 6.5 years, including post-treatment survival follow up period. Serious and Other Adverse Events: from first dose of study treatment until 30 days after last dose up to approx. 6.5 years
Description: All-cause mortality: reported for all randomized participants regardless of whether the assigned study treatment was received. Deaths in post-treatment survival follow (more than 30 days after last dose) are reported separately and are not considered AEs.
  Serious and Other Adverse Events: reported for all randomized participants who received any amount of study treatment
Groups:
- Alpelisib + Fulvestrant; Placebo + Fulvestrant: All-cause mortality from randomization until 30 days after last dose. Adverse Events from first dose until 30 days after last dose.
- Alpelisib + Fulvestrant (Post-treatment Survival Follow-up); Placebo + Fulvestrant (Post-treatment Survival Follow-up): Deaths collected in the post- treatment survival follow-up period (starting from day 31 after last dose). No AEs were collected during this period
Arm/Group | Alpelisib + Fulvestrant | Placebo + Fulvestrant | Alpelisib + Fulvestrant (Post-treatment Survival Follow-up) | Placebo + Fulvestrant (Post-treatment Survival Follow-up)
All-Cause Mortality (participants affected / at risk) | 9/284 | 12/288 | 151/275 | 156/275
Serious Adverse Events (participants affected / at risk) | 110/284 | 54/287 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 280/284 | 244/287 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alpelisib + Fulvestrant (N=284) | Placebo + Fulvestrant (N=287) | Alpelisib + Fulvestrant (Post-treatment Survival Follow-up) (N=0) | Placebo + Fulvestrant (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 6 | 0 | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | NA | NA
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0 | NA | NA
Angina pectoris (Cardiac disorders) | 0 | 1 | NA | NA
Arteriospasm coronary (Cardiac disorders) | 1 | 0 | NA | NA
Atrial fibrillation (Cardiac disorders) | 1 | 1 | NA | NA
Bradycardia (Cardiac disorders) | 1 | 0 | NA | NA
Cardiac arrest (Cardiac disorders) | 1 | 0 | NA | NA
Cardiac failure (Cardiac disorders) | 0 | 1 | NA | NA
Myocardial infarction (Cardiac disorders) | 0 | 1 | NA | NA
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | NA | NA
Pericardial effusion (Cardiac disorders) | 0 | 1 | NA | NA
Sinus tachycardia (Cardiac disorders) | 0 | 1 | NA | NA
Supraventricular tachycardia (Cardiac disorders) | 2 | 0 | NA | NA
Cataract (Eye disorders) | 0 | 2 | NA | NA
Abdominal pain (Gastrointestinal disorders) | 6 | 2 | NA | NA
Colitis (Gastrointestinal disorders) | 2 | 1 | NA | NA
Constipation (Gastrointestinal disorders) | 0 | 1 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 9 | 0 | NA | NA
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | NA | NA
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | NA | NA
Gallstone ileus (Gastrointestinal disorders) | 0 | 1 | NA | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | NA | NA
Ileus (Gastrointestinal disorders) | 1 | 0 | NA | NA
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | NA | NA
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | NA | NA
Melaena (Gastrointestinal disorders) | 1 | 0 | NA | NA
Nausea (Gastrointestinal disorders) | 5 | 2 | NA | NA
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | NA | NA
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | NA | NA
Stomatitis (Gastrointestinal disorders) | 4 | 0 | NA | NA
Subileus (Gastrointestinal disorders) | 0 | 1 | NA | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | NA | NA
Vomiting (Gastrointestinal disorders) | 5 | 3 | NA | NA
Adverse drug reaction (General disorders) | 1 | 0 | NA | NA
Asthenia (General disorders) | 1 | 0 | NA | NA
Chest discomfort (General disorders) | 1 | 0 | NA | NA
Chest pain (General disorders) | 1 | 0 | NA | NA
Fatigue (General disorders) | 1 | 0 | NA | NA
General physical health deterioration (General disorders) | 2 | 0 | NA | NA
Malaise (General disorders) | 1 | 0 | NA | NA
Mucosal inflammation (General disorders) | 3 | 0 | NA | NA
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | NA | NA
Pyrexia (General disorders) | 4 | 0 | NA | NA
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | NA | NA
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | NA | NA
Anaphylactic reaction (Immune system disorders) | 1 | 0 | NA | NA
Hypersensitivity (Immune system disorders) | 3 | 0 | NA | NA
Abdominal infection (Infections and infestations) | 1 | 0 | NA | NA
Abscess jaw (Infections and infestations) | 1 | 0 | NA | NA
Appendicitis (Infections and infestations) | 0 | 1 | NA | NA
Bacteraemia (Infections and infestations) | 1 | 0 | NA | NA
COVID-19 (Infections and infestations) | 1 | 0 | NA | NA
Cellulitis (Infections and infestations) | 2 | 2 | NA | NA
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 1 | 0 | NA | NA
Erysipelas (Infections and infestations) | 1 | 0 | NA | NA
Herpes zoster (Infections and infestations) | 1 | 0 | NA | NA
Mediastinitis (Infections and infestations) | 0 | 1 | NA | NA
Peritonsillar abscess (Infections and infestations) | 1 | 0 | NA | NA
Pneumonia (Infections and infestations) | 3 | 6 | NA | NA
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | NA | NA
Pyelonephritis (Infections and infestations) | 1 | 1 | NA | NA
Pyelonephritis acute (Infections and infestations) | 1 | 0 | NA | NA
Respiratory tract infection (Infections and infestations) | 1 | 1 | NA | NA
Septic shock (Infections and infestations) | 0 | 1 | NA | NA
Skin infection (Infections and infestations) | 0 | 1 | NA | NA
Urinary tract infection (Infections and infestations) | 2 | 3 | NA | NA
Urosepsis (Infections and infestations) | 1 | 0 | NA | NA
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1 | NA | NA
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Radiation proctitis (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1 | NA | NA
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Alanine aminotransferase increased (Investigations) | 1 | 0 | NA | NA
Aspartate aminotransferase increased (Investigations) | 1 | 0 | NA | NA
Blood bilirubin increased (Investigations) | 0 | 1 | NA | NA
Blood creatinine increased (Investigations) | 2 | 0 | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | NA | NA
Haemoglobin decreased (Investigations) | 1 | 0 | NA | NA
Hepatic enzyme increased (Investigations) | 1 | 0 | NA | NA
Lipase increased (Investigations) | 1 | 0 | NA | NA
Weight decreased (Investigations) | 1 | 0 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | NA | NA
Dehydration (Metabolism and nutrition disorders) | 3 | 3 | NA | NA
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0 | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 28 | 0 | NA | NA
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | NA | NA
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 9 | 2 | NA | NA
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Altered state of consciousness (Nervous system disorders) | 0 | 1 | NA | NA
Brain oedema (Nervous system disorders) | 2 | 0 | NA | NA
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | NA | NA
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | NA | NA
Headache (Nervous system disorders) | 1 | 0 | NA | NA
Motor dysfunction (Nervous system disorders) | 0 | 1 | NA | NA
Seizure (Nervous system disorders) | 1 | 0 | NA | NA
Spinal cord compression (Nervous system disorders) | 0 | 2 | NA | NA
Syncope (Nervous system disorders) | 1 | 0 | NA | NA
Bipolar disorder (Psychiatric disorders) | 1 | 0 | NA | NA
Suicide attempt (Psychiatric disorders) | 0 | 1 | NA | NA
Acute kidney injury (Renal and urinary disorders) | 6 | 1 | NA | NA
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | NA | NA
Renal failure (Renal and urinary disorders) | 2 | 0 | NA | NA
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | NA | NA
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | NA | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | NA | NA
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | NA | NA
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 | 0 | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 5 | 0 | NA | NA
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | NA | NA
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA
Deep vein thrombosis (Vascular disorders) | 1 | 0 | NA | NA
Hypertension (Vascular disorders) | 1 | 0 | NA | NA
Thrombosis (Vascular disorders) | 0 | 1 | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alpelisib + Fulvestrant (N=284) | Placebo + Fulvestrant (N=287) | Alpelisib + Fulvestrant (Post-treatment Survival Follow-up) (N=0) | Placebo + Fulvestrant (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 29 | 20 | NA | NA
Vision blurred (Eye disorders) | 15 | 2 | NA | NA
Abdominal pain (Gastrointestinal disorders) | 33 | 20 | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 19 | 13 | NA | NA
Constipation (Gastrointestinal disorders) | 25 | 37 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 167 | 48 | NA | NA
Dry mouth (Gastrointestinal disorders) | 30 | 13 | NA | NA
Dyspepsia (Gastrointestinal disorders) | 32 | 17 | NA | NA
Nausea (Gastrointestinal disorders) | 133 | 64 | NA | NA
Stomatitis (Gastrointestinal disorders) | 70 | 20 | NA | NA
Vomiting (Gastrointestinal disorders) | 80 | 27 | NA | NA
Asthenia (General disorders) | 64 | 40 | NA | NA
Fatigue (General disorders) | 73 | 51 | NA | NA
Mucosal inflammation (General disorders) | 53 | 4 | NA | NA
Oedema peripheral (General disorders) | 46 | 14 | NA | NA
Pyrexia (General disorders) | 47 | 16 | NA | NA
Nasopharyngitis (Infections and infestations) | 24 | 26 | NA | NA
Upper respiratory tract infection (Infections and infestations) | 15 | 19 | NA | NA
Urinary tract infection (Infections and infestations) | 28 | 13 | NA | NA
Alanine aminotransferase increased (Investigations) | 28 | 18 | NA | NA
Aspartate aminotransferase increased (Investigations) | 32 | 18 | NA | NA
Blood creatinine increased (Investigations) | 36 | 4 | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 28 | 23 | NA | NA
Lipase increased (Investigations) | 21 | 12 | NA | NA
Weight decreased (Investigations) | 79 | 7 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 103 | 30 | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 182 | 27 | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 25 | 5 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 44 | 56 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 44 | 43 | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 14 | 19 | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 23 | 12 | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 20 | 9 | NA | NA
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 15 | 3 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 29 | 24 | NA | NA
Dizziness (Nervous system disorders) | 27 | 20 | NA | NA
Dysgeusia (Nervous system disorders) | 39 | 8 | NA | NA
Headache (Nervous system disorders) | 53 | 38 | NA | NA
Insomnia (Psychiatric disorders) | 22 | 12 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 28 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 | 32 | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 58 | 7 | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 44 | 10 | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 19 | 2 | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 54 | 19 | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 101 | 20 | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 39 | 4 | NA | NA
Hot flush (Vascular disorders) | 9 | 19 | NA | NA
Hypertension (Vascular disorders) | 29 | 15 | NA | NA
Lymphoedema (Vascular disorders) | 17 | 6 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT02437318/Prot_002.pdf
  • Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT02437318/SAP_003.pdf